CLINICAL TRIAL: NCT04462549
Title: Improving Health Outcomes Following Traumatic Brain Injury Through Building a TBI-informed System of Services and Supports and Resource Facilitation
Brief Title: Improving Health Outcomes With Resource Facilitation
Acronym: ACL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rehabilitation Hospital of Indiana (Other)
Responsible Party: Principal Investigator, Devan Parrott, Director and Biostatistician, Rehabilitation Hospital of Indiana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1811467577
Record Dates: First submitted 2019-08-08; First posted 2020-07-08 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Traumatic Brain Injury; Rehabilitation; Intervention
Keywords: Resource Facilitation
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial 100 subjects who will participate in this study will be randomly assigned to the Resource Facilitation Group. These subjects will receive resource facilitation services in addition to their regular rehabilitation follow-up services, and 50 subjects who will participate in this study will be randomly assigned to the Regular Follow-up Group, who will only receive their regular rehabilitation follow-up services/standard of care. Randomization will be generated within RedCap.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resource Facilitation (Experimental): This group is receiving Resource Facilitation
  Interventions: Behavioral: Resource Facilitation
- Control (No Intervention): Not receiving Resource Facilitation

INTERVENTIONS:
Behavioral: Resource Facilitation — RF involves working one on one with a brain injury specialist. This specialist is called a "Resource Facilitator" and works with clients to help set and achieve their own goals along with a team of professionals that specialize in this kind of injury. This may include brain injury education, family education, needs assessments, and service identification.
  Arms: Resource Facilitation

SUMMARY:
The purpose of this research is to test a service the investigators of the study believe may increase quality of life after brain injury and reduce the level of disability that might be associated with that injury.

This intervention is called "Resource Facilitation" and involves working one on one with a brain injury specialist. This specialist is called a "Resource Facilitator" and will work with participants to help set and achieve their own goals along with a team of professionals that specialize in this kind of injury. If randomly assigned to the Resource Facilitation group, participants will receive Resource Facilitation free of charge. If not, they will be assigned to a control group and will not receive the intervention. However, both groups will receive calls every three months. During these calls, a research assistant will collect data about each participant's recovery and progress. If assigned to the Resource Facilitation group, participants may also receive study information in the mail if research assistants are unable to reach participants via telephone.

DETAILED DESCRIPTION:
Approximately 2.5 million people are hospitalized each year for traumatic brain injury (TBI) in the United States, according to the Centers for Disease Control and Prevention. The Indiana State Department of Health (ISDH) found in 2013 that more than 50,000 Hoosiers suffered a traumatic brain injury (TBI). Further, the prevalence of TBI-related disability in Indiana was found to be 66,410. These findings clearly indicate that Indiana has a significant health care and social burden associated with TBI.

To date, investigators have made substantial progress through our previous TBI HRSA grants in the development and evaluation of the RF model as applied to vocational rehabilitation outcomes. However, there are many people in Indiana who do not have access to these services. Further, TBI is now recognized to be a chronic health condition, and investigators have not implemented Resource Facilitation (RF) to improve or stabilize health outcomes.

Through our 2009-2014 HRSA TBI grant, investigators became interested in the RF model, but noted the absence of empirical outcome data to support its effectiveness. To address this need, investigators conducted the first randomized controlled trial of RF with 22 participants who were recruited while they were still in acute brain injury rehabilitation, and were, on average, approximately 3 months post-injury. The participants were randomized to RF or a treatment as usual control group. After six months, it was found that 64% of the RF treatment group was successful at returning to competitive employment as compared to 36% of the control group (Wald-Wolfkowitz z = -3.277, p < .0001). While it was found that both groups had reduced level of disability at follow-up (F = 60.65, p < .0001), it was also found that the interaction for groups and time was significant (F = 9.11, p = .007) indicating that the participants who received RF were significantly less disabled at follow-up as compared to the control participants.

These findings were replicated in a larger randomized controlled trial that studied 44 participants with acquired brain injury that were again approximately 2-3 months post-injury. Participants were randomized to 12 months of RF or a treatment as usual control group. The results again demonstrated a significant advantage for the RF group (69%) for both rate of return to work as compared to the control group (50%) and how quickly they returned to work. Using a logistic regression, investigators found that group assignment was a significant predictor of vocational outcome (Wald = 4.91, p= .027) and RF participants were found to be seven times more likely to return to productive community-based work as compared to controls (95% confidence interval, 1.25-39.15). The evidence supporting the efficacy of RF seemed sufficient to support a clinical trial to examine effectiveness.

Based on these two publications, Indiana Vocational Rehabilitation supported a prospective clinical cohort study of the effectiveness of RF. In this study, investigators provided RF to 210 clients of Indiana Vocational Rehabilitation and compared their vocational outcomes to the participants in the control groups in our two previous randomized controlled trials. In contrast to our randomized controlled trials, these participants who received RF were almost 10 years post-injury. Of the 210 participants in the RF treatment group, 69% (n=145) successfully returned to competitive work. Six of these 145 successful outcomes were for participants that had a goal of return to post-high school education. Investigators compared these outcomes for the RF cohort with the outcomes attained by the control groups from our two previous randomized controlled trials and found that 48% (n=16) of the control participants successfully returned to paid employment. The difference between the two groups revealed a significant advantage for the RF group (Χ2(1)=5.39, p = .018). These results certainly provided evidence for the effectiveness of RF for helping people get back to work after acquired brain injury in a cohort referred to us by Indiana Vocational Rehabilitation.

Based on the success of our HRSA TBI grants and the results from the first two randomized controlled trials and the prospective clinical cohort study, Indiana Vocational Rehabilitation decided to support RF for any person with a brain injury and who qualified for services in 2014, and RF was made available throughout the state of Indiana by 2015. Today, approximately 350 individuals with acquired brain injury are receiving RF at any one time. However, it is quite noteworthy that investigators had more than 700 referrals from the community for RF, the vast majority of which will not qualify for Indiana Vocational Rehabilitation services. It is for these reasons that in Indiana, investigators need to expand access to RF to promote optimal health outcomes and decrease disability associated with TBI.

ELIGIBILITY:
Inclusion Criteria:

-Documented TBI (if one or more of the following criteria apply: Loss of consciousness of 30 minutes or more Post-traumatic anterograde amnesia of 24 hours or more Worst Glasgow Coma Scale full score in first 24 hours < 13 (unless invalidataed upon review, e.g., attributable to intoxication, sedation, systemic shock)

* One or more of the following present: Intracerebral hematoma, Subdural hematoma, Epidural hematoma, Cerebral contusion, Hemorrhagic contusion, Penetrating TBI (dura penetrated), Subarachnoid hemorrhage, Brain stem injury
* Resides in one of the following counties: Vigo, Clay, Parke, Vermillion, Fountain, Warren, Tippecanoe, Montgomery, Putnam, Owen, Monroe, Brown, Morgan, Hendricks, Boone, Clinton, Howard, Tipton, Hamilton, Marion, Johnson, Bartholomew, Shelby, Hancock, Madison, Delaware, Henry, Rush, Decatur, Randolph, Wayne, Fayette, Union, or Franklin
* Age older than 17

Exclusion Criteria:

* From or going to jail or prison following injury
* Anyone with pre-existing progressive CNS disorder (this does not include previous TBI or stroke, for example)
* Being discharged from Acute Hospital LTAC
* Anyone who cannot interact with the environment
* Unable to follow commands

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-01-13 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Patient reported outcome measurement information system (PROMIS): Health Related Quality of Life (HRQL) | 3 months, 6 months, 9 months, 12 months, 15 months
  The PROMIS subscales are patient reported outcome measures available through NIH with excellent reliability and validity. The HRQL construct includes the following subscales: Depression, Anxiety, Physical Functioning, Social Participation, Pain Interference, Pain Intensity, Sleep Disturbance, and Fatigue. Higher scores suggest greater quality of life in the subscales above.
Change in Quality of Life after Brain Injury (QOLIBRI) | 3 months, 6 months, 9 months, 12 months, 15 months
  This measures quality of life (QOL) symptoms unique to the brain injury population. Participants rate each statement from 1 (Not at all) to 5 (Very). Higher scores represent greater quality of life after experiencing brain injury
Change in Charlson Comorbidity List | 3 months, 6 months, 9 months, 12 months, 15 months
  This list is a well-established list of comorbidities to chronic diseases based on the International Classification of Diseases (ICD) codes. The final score is a sum of weights associated with each comorbidity reported with higher scores representing an increased likelihood for resource use/mortality.
Change in Traumatic Brain Injury (TBI) Symptom and Functional Status Checklist | 3 months, 6 months, 9 months, 12 months, 15 months
  This symptom checklist is not a normed, validated checklist, but rather a list of common brain injury symptoms observed both clinically and well-documented in the literature. This list is being piloted in this study but will provide a simple quantifier for TBI symptoms reported per patient. This form also includes key demographic information and variables that may change during the course of treatment (contact information, insurance, marital status, list of medications) that will not be considered primary outcomes.
Change in Mayo-Portland Adaptability Inventory - IV (MPAI-4) | 3 months, 6 months, 9 months, 12 months, 15 months
  This measure is designed for outcome measurement after acquired brain injury in the post acute stage of recovery. The MPAI-4 is the product of 15 years of development using item response and classic psychometric theory and has established concurrent, construct, and predictive validity. There is a total score and subscale scores for Ability, Adjustment, and Participation Greater scores represent greater need in the subscales mentioned before.

SECONDARY OUTCOMES:
Change in Vocational Independence Scale - Revised (VIS-R) | up to two weeks, 3 months, 6 months, 9 months, 12 months, 15 months
  This was created to measure the level of employment based on independence and hours worked with/without supervision. This measure was revised by the study PIs to include academic attainment. On a scale of 1-5, individuals select which statement best matches their vocational/educational status.
Change in Survey of Unmet Needs and Services Utilized (SUNSU) | 3 months, 6 months, 9 months, 12 months, 15 months
  This measure was designed to assess both the usage of services as well as desired services within the brain injury community. The measure shows strong internal consistency when compared to other needs assessments in the brain injury population and results in two scores: the number of items currently received (met needs) and number of items desired (unmet needs).

OTHER OUTCOMES:
Change in Headache Impact Test 6 (HIT6) | Up to 2 weeks, 3 months, 6 months, 9 months, 12 months, 15 months
  This is a well validated measure of impact of episodic and chronic migraines on social functioning, role functioning, vitality, cognitive functioning and psychological distress.
Orientation Log (O-Log) | Up to 2 weeks
  This measures patient orientation to time and place in populations with potential impairments to orientation and confusion. This measure will provide a brief objective measure of confusion and will be used as a covariate when interpreting other outcome measures.
Change in Behavioral Rating Inventory of Executive Function-Adult Version (Brief-A) | 3 months, 6 months, 9 months, 12 months, 15 months
  consists of 75 items reflecting overall executive function. Scores can be broken down into nine subscales as well as two summary index scales. Participants rate how much they experience each statement on a scale of Never, Sometimes, or Often.

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabilitation Hospital of Indiana, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No